CLINICAL TRIAL: NCT00879034
Title: A Phase II Pilot Study of Zoledronic Acid, Pravastatin, and Lonafarnib (SCH66336) for Patients With Hutchinson-Gilford Progeria Syndrome (HGPS) and Progeroid Laminopathies
Brief Title: A Study of Zoledronic Acid, Pravastatin, and Lonafarnib for Patients With Progeria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Schering-Plough (Industry)
Responsible Party: Principal Investigator, Monica E. Kleinman, Critical Care, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-02-0074; P06087 (Other: Schering-Plough)
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Progeria; Hutchinson-Gilford Syndrome
Keywords: Hutchinson-Gilford Progeria Syndrome; HGPS; Progeria; FTI; Farnesyltransferase Inhibitor; Lonafarnib; Zoledronic Acid; Pravastatin
MeSH Terms: conditions — Progeria | interventions — lonafarnib; Zoledronic Acid; Pravastatin

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zoledronic Acid,Pravastatin,and Lonafarnib (Experimental): Lonafarnib;Zoledronic acid;Pravastatin
  Interventions: Drug: Lonafarnib; Drug: Zoledronic Acid; Drug: Pravastatin

INTERVENTIONS:
Drug: Lonafarnib — Lonafarnib capsules are to be orally administered twice per day approximately every 12 hours. Lonafarnib dosing will begin at 150 mg/m2 by mouth twice daily. Dose levels are 150, 115, 90 and 70 mg/m2. Patients experiencing significant drug related grade 3 or 4 toxicity and not responding to therapy interruption or supportive care measures will be dose reduced by one dose level.
  Other Names: Sarasar, SCH 66336
Drug: Zoledronic Acid — Zoledronic acid will be administered intravenously at week one of this treatment trial. Week one administration will consist of one infusion over a 30 minute period, 0.0125 mg/kg body weight.
  Other Names: Zometa, Reclast
Drug: Pravastatin — Pravastatin will begin at 5 mg by mouth once daily for children weighing less than 10 kg, and 10 mg by mouth once daily for children weighing 10 kg or greater.
  Other Names: Pravachol

SUMMARY:
This is an open label single arm feasibility trial. A combination of two oral agents (pravastatin and lonafarnib) and one intravenous (IV) agent (zoledronic acid) will be administered at doses and schedule currently applied in pediatrics. These agents all target farnesylation pathways at different points. Our goal is to inhibit farnesylation of abnormal lamin, the disease-causing protein in Hutchinson-Gilford Progeria Syndrome and progeroid laminopathies (henceforth "progeria"). The drugs will include the intravenous bisphosphonate zoledronic acid, oral HMG co-reductase inhibitor pravastatin and the oral farnesyltransferase inhibitor (FTI) lonafarnib (SCH 66336). Patients with genetically confirmed progeria will be eligible for this protocol. Treatment will be initiated for 4 weeks duration and may be extended depending on tolerability. This study will assess the feasibility of this treatment regimen in the first 4 weeks. If tolerated for 4 weeks, patients can be treated with this regimen for up to 6 months.

DETAILED DESCRIPTION:
Progerias are rare "premature aging" diseases in which children die of severe atherosclerosis leading to strokes and heart attacks. It is a multisystem disease with objective clinical markers for disease progression. These include abnormalities in growth and body composition, bone mineral density, join function, endocrine function, alopecia, and vascular disease. There is currently no therapy proven effective for any of the progressive and deleterious aspects of this disorder.

Progeria is caused by a gene defect in the gene LMNA, coding for the nuclear protein lamin A. Lamin A is normally expressed by most differentiated cells, and requires posttranslational farnesylation to incorporate into the nuclear membrane. This trial proposes to use three agents (zoledronic acid, pravastatin, and lonafarnib) to inhibit farnesylation of abnormal lamin, the disease causing protein in Progeria. The primary objective of this study is to evaluate the feasibility of administering intravenous zoledronic acid, oral pravastatin and oral lonafarnib, to patients wtih Progeria for a minimum of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Genetic Diagnosis: All patients must have confirmatory mutational analysis showing mutation in the lamin A gene.
* Patients must display clinical signs of progeria as per the clinical trial team.
* Patients must be willing and able to come to Boston for appropriate studies and examinations at initiation of study and at week 4 of study.
* Patient must have adequate organ and marrow function as defined by study parameters

Exclusion Criteria:

* Other than the drugs used in this protocol, other drugs targeted to treat Progeria are excluded. Drugs to treat symptoms of Progeria are permitted.
* Patients must not be taking medications that significantly affect the metabolism of lonafarnib at the time they start lonafarnib.
* Patient must have no uncontrolled infection.
* Subjects who have known or suspected hypersensitivity to any of the excipients included in the formulation should not be treated.
* Patients must not be pregnancy of breast-feeding. Female patients of childbearing potential must have negative serum or urine pregnancy test. Male and female patients of reproductive potential must agree to use a medically accepted form of birth control while on study and up to 10 weeks after treatment. It is permissible for female patients to take oral contraceptives or other hormonal methods while receiving treatment with lonafarnib.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Kieran, MD, PhD, Study Chair — Dana-Farber Cancer Institute; Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gordon LB, Massaro J, D'Agostino RB Sr, Campbell SE, Brazier J, Brown WT, Kleinman ME, Kieran MW; Progeria Clinical Trials Collaborative. Impact of farnesylation inhibitors on survival in Hutchinson-Gilford progeria syndrome. Circulation. 2014 Jul 1;130(1):27-34. doi: 10.1161/CIRCULATIONAHA.113.008285. Epub 2014 May 2. PMID 24795390
- [Result] Gordon LB, Kleinman ME, Massaro J, D'Agostino RB Sr, Shappell H, Gerhard-Herman M, Smoot LB, Gordon CM, Cleveland RH, Nazarian A, Snyder BD, Ullrich NJ, Silvera VM, Liang MG, Quinn N, Miller DT, Huh SY, Dowton AA, Littlefield K, Greer MM, Kieran MW. Clinical Trial of the Protein Farnesylation Inhibitors Lonafarnib, Pravastatin, and Zoledronic Acid in Children With Hutchinson-Gilford Progeria Syndrome. Circulation. 2016 Jul 12;134(2):114-25. doi: 10.1161/CIRCULATIONAHA.116.022188. PMID 27400896
- [Derived] Gordon LB, Norris W, Hamren S, Goodson R, LeClair J, Massaro J, Lyass A, D'Agostino RB Sr, Tuminelli K, Kieran MW, Kleinman ME. Plasma Progerin in Patients With Hutchinson-Gilford Progeria Syndrome: Immunoassay Development and Clinical Evaluation. Circulation. 2023 Jun 6;147(23):1734-1744. doi: 10.1161/CIRCULATIONAHA.122.060002. Epub 2023 Mar 15. PMID 36919608
- [Derived] Fisher MJ, Avery RA, Allen JC, Ardern-Holmes SL, Bilaniuk LT, Ferner RE, Gutmann DH, Listernick R, Martin S, Ullrich NJ, Liu GT; REiNS International Collaboration. Functional outcome measures for NF1-associated optic pathway glioma clinical trials. Neurology. 2013 Nov 19;81(21 Suppl 1):S15-24. doi: 10.1212/01.wnl.0000435745.95155.b8. PMID 24249802
- See also: Progeria Research Foundation — http://www.progeriaresearch.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 patients with classic HGPS from the United States were enrolled in March 2009 at Boston Children's Hospital. 1 additional patient had nonclassic mutations.
Pre-assignment Details: All patients screened to participate in study were consented onto the study as planned.
Groups:
- Zoledronic Acid, Pravastatin, and Lonafarnib: Lonafarnib capsules are to be orally administered twice per day approximately every 12 hours. Lonafarnib dosing will begin at 150 mg/m2 by mouth twice daily. Dose levels are 150, 115, 90 and 70 mg/m2. Patients experiencing significant drug related grade 3 or 4 toxicity and not responding to therapy interruption or supportive care measures will be dose reduced by one dose level. Zoledronic acid will be administered intravenously at week one of this treatment trial. Week one administration will consist of one infusion over a 30 minute period, 0.0125 mg/kg body weight. Pravastatin will begin at 5 mg by mouth once daily for children weighing less than 10 kg, and 10 mg by mouth once daily for children weighing 10 kg or greater.
Period: Overall Study
Arm/Group | Zoledronic Acid, Pravastatin, and Lonafarnib
Started | 5
Received Treatment (One patient did not receive a zoledronic acid infusion during study.) | 4
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zoledronic Acid, Pravastatin, and Lonafarnib
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Study is to Evaluate the Feasibility of Administering Intravenous Zoledronic Acid, Oral Pravastatin and Oral Lonafarnib, to Patients With Progeria for a Minimum of 4 Weeks
Description: Feasibility was assessed by determining the number of participants with adverse events occurring over the course of the 4 week study.
Time Frame: 4 weeks
Population: Results are reported for the 5 patients who completed the 4 weeks of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid, Pravastatin, and Lonafarnib
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: To Describe Any Acute and Chronic Toxicities Associated With Treating Progeria Patients With the Combination of Zoledronic Acid, Pravastatin and Lonafarnib
Description: Number of participants with acute and chronic toxicities associated with treating progeria patients with the combination of zoledronic acid, pravastatin and lonafarnib
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid, Pravastatin, and Lonafarnib
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: To Investigate Which Clinical and Laboratory Studies Are Needed to Monitor or Alter Therapy to Prevent Unacceptable Toxicity
Description: The number of participants with abnormal CBC w/diff panel, LFTs, renal functions and lipid panels.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid, Pravastatin, and Lonafarnib
Number analyzed (Participants) | 5
Participants | 0

4. Secondary Outcome: To Assess the Pharmacokinetics of Lonafarnib in Patients With Progeria.
Time Frame: 4 weeks
Population: This data was not collected for this feasibility study. Pharmacokinetics assessment of lonafarnib in these 5 patients was analyzed at the end of a different protocol, NCT00916747.
Arm/Group | Zoledronic Acid, Pravastatin, and Lonafarnib
Number analyzed (Participants) | 0

5. Secondary Outcome: To Assay for the Inhibition of HDJ-2 Farnesylation in Peripheral Blood Leukocytes (PBL)
Time Frame: 4 weeks
Population: This data was not collected for this feasibility study. HDJ-2 assessment in these 5 patients was analyzed at the end of a different protocol, NCT00916747.
Arm/Group | Zoledronic Acid, Pravastatin, and Lonafarnib
Number analyzed (Participants) | 0

6. Secondary Outcome: To Obtain Baseline Clinical and Laboratory Data so That Longer-term Measures of Efficacy Will be Achievable if Treatment Continues Beyond the 4-week Feasibility Study Period.
Description: The number of participants from whom baseline clinical and Laboratory data was obtained.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid, Pravastatin, and Lonafarnib
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: Up to 4 weeks. Assessed at week 0 and week 4.
Arm/Group | Zoledronic Acid, Pravastatin, and Lonafarnib
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
This was an open label clinical trial on a very rare disease population. Patient numbers are small, though 5 participants represents a small but significant portion of the world's population of children with HGPS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No